CLINICAL TRIAL: NCT00151554
Title: Reducing ICU Related Anxiety Through a Structured Information Program. A Randomized Controlled Clinical Trial
Brief Title: Reducing Intensive Care Unit (ICU) Related Anxiety Through a Structured Information Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Pflegeverbund Mitte-Süd (Unknown); Stabstelle Pflegeforschung (Unknown); Institut für Theoretische Chirurgie (Unknown); Klinik für Herzchirurgie (Unknown); Klinik für VTG-Chirurgie (Unknown)
Responsible Party: Dr. Thomas R. Neubert, Philipps University Marburg Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PflegeverbundMarburg2; BMBF grant 01GT0303
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-07

CONDITIONS: Heart Diseases
Keywords: Anxiety; Intensive Care Unit (ICU); Preoperative Information; Randomized Controlled Trial (RCT); Chronic heart disease
MeSH Terms: conditions — Heart Diseases; Anxiety Disorders

ARMS (2):
- Control group (No Intervention)
- Intervention group (Experimental)
  Interventions: Behavioral: ICU-specific information program

INTERVENTIONS:
Behavioral: ICU-specific information program — The intervention group receives a standardized information program with specific procedural, sensory and coping information about the ICU in addition to standard information given by surgeons and anesthetists.
  Arms: Intervention group

SUMMARY:
According to current evidence and psychological theorizing, the provision of information seems to be a promising way to reduce the anxiety of patients that is related to their scheduled ICU stay. An ICU-specific information program will be investigated in a randomized controlled clinical trial involving 120 patients undergoing elective open heart surgery and 20 patients undergoing abdominal surgery. It is expected that the patients in the test group will experience less anxiety and ICU related discomfort than patients in the control group.

DETAILED DESCRIPTION:
Objective: According to current evidence and psychological theorizing the provision of information seems to be a promising way to reduce anxiety of patients. In the case of surgical patients, admission to the intensive care unit (ICU) is strongly associated with uncertainty, unpredictability and anxiety for the patient. Thus, ICU-specific information could have a high clinical impact. For this reason this study will evaluate the efficacy of an ICU-specific information program for patients who undergo elective cardiac, abdominal or thoracic surgery and are scheduled for ICU stay.

Methods: The trial is designed as a prospective randomized controlled trial including an intervention and a control group. The control group receives the standard preparation currently conducted by surgeons and anesthesists. The intervention group additionally receives a standardized information program with specific procedural, sensory and coping information about the ICU. In addition the moderating effect of certain personality characteristics (need for cognition, high trait anxiety) will be investigated to identify groups of patients who benefit most from the information program.

Expected Results: A clinically relevant difference in anxiety and unpleasant experiences related to the ICU is expected after discharge from the ICU. Power calculation (alpha = 0.05; beta = 0.20; delta = 8.50 score points) resulted in a required sample size of N = 120 cardiac surgical patients (n = 60 vs. n = 60). Furthermore, N = 20 abdominal or thoracic surgical patients will be recruited (n = 10 vs. n = 10).

Conclusion: The proposed study promises to strengthen evidence on the effects of a specific, concise information program and thus should contribute to evidence based nursing (EBN).

ELIGIBILITY:
Inclusion Criteria:

* Elective open heart or abdominal surgery including scheduled ICU stay
* Informed consent

Exclusion Criteria:

* Elective surgery without ICU stay
* Informed consent denied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2005-02; Primary Completion 2006-09 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Patient self-reported anxiety | after admission on standard ward
ICU related discomfort | after admission on standard ward

SECONDARY OUTCOMES:
Objective health status parameters | postoperative phase of hospital stay
Overall satisfaction with care | 3 months after discharge
Quality of life | 3 months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Neubert, PhD, Principal Investigator — Stabstelle Pflegeforschung, Universitätsklinikum Marburg
Locations (1):
- University Hospital Marburg, Marburg, Hesse, Germany

REFERENCES:
- [Background] Berg A, Fleischer S, Koller M, Neubert TR. Preoperative information for ICU patients to reduce anxiety during and after the ICU-stay: protocol of a randomized controlled trial [NCT00151554]. BMC Nurs. 2006 Mar 8;5:4. doi: 10.1186/1472-6955-5-4. PMID 16524468